CLINICAL TRIAL: NCT01693861
Title: Molecularly Imprinted Polymer Sensors of Modified Nucleosides for Non-invasive Monitoring of Cancer Therapy : Effect of Chemotherapy on Cancerous Proliferation Based on the Dynamic Excretion of Urinary Nucleosides.
Brief Title: "Cancersensor" Chemotherapy
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-59; 2012-A00168-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-09-07; First posted 2012-09-26 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2016-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal; Cancer; Metastatic; Chronotherapy; Urine; Nucleosides; Chemotherapy; Treated with chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and exfoliated oral mucosa cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with metastatic colorectal cancer treated with chemotherapy

SUMMARY:
Observational, non randomized study aimed at measuring the effect of chemotherapy in the urinary concentrations of physiological modified nucleosides in 30 patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed metastatic colorectal cancer;
* 0 to 3 prior chemotherapy lines;
* Signed informed consent;
* Good understanding of the protocol and of the follow-up;
* Estimated life expectancy exceeding 3 months;
* At least one measurable metastatic lesion (RECIST criteria);
* Performance Status (WHO) of 0 to 2;
* Good haematological, hepatic and renal functions.

Exclusion Criteria:

* More than 2 surgical resections of metastases from colorectal cancer;
* Poor performance status (>2);
* Poor haematological, hepatic or renal functions;
* Uncontrolled chronic disease;
* Serious unhealed wound, ulcer or fracture within the previous month;
* Clinical or laboratory finding suggesting possible abnormalities in nucleosides urinary excretion;
* Pregnancy or breast-feeding during the previous month;
* Transmeridian trip of more than 4 time zones within the prior 2 weeks;
* Person with legal restriction to participate into clinical research, according to the current law in France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer treated at the Department of Medical Oncology of Paul Brousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Effect of chemotherapy on urinary excretion of modified nucleosides | 17 days
  1 urine sample per day 3 days before and 14 days after beginning of chemotherapy Measurement of modified nucleosides, cortisol and 6-sulfatoxymelatonin concentration
  1 saliva sample : Measurement of Clock genes polymorphisms expression

OTHER OUTCOMES:
Identification of modified nucleosides as biomarkers for colorectal cancer | 17 days
  Measurement of modified nucleosides, cortisol and 6-sulfatoxymelatonin concentration in urine samples before and after chemotherapy
  1 saliva sample Measurement of Clock genes polymorphisms expression

CONTACTS AND LOCATIONS:
Overall Officials: Francis Lévi, MD PhD, Principal Investigator — INSERM CNRS AP-HP Université Paris Sud
Locations (1):
- Paul Brousse Hospital, Villejuif, France

REFERENCES:
- [Result] Dulong S, Huang Q, Innominato PF, Karaboue A, Bouchahda M, Pruvost A, Theodoro F, Agrofoglio LA, Adam R, Finkenstadt B, Levi F. Circadian and chemotherapy-related changes in urinary modified nucleosides excretion in patients with metastatic colorectal cancer. Sci Rep. 2021 Dec 14;11(1):24015. doi: 10.1038/s41598-021-03247-2. PMID 34907230